CLINICAL TRIAL: NCT01474083
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group, Multiple-Dose Study Assessing the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of GK1-399 in Patients With Type 2 Diabetes Mellitus
Brief Title: A 6 Week Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of GK1-399 in Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: vTv Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GK1-MS-201
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GK1-399, low dose (Experimental)
  Interventions: Drug: GK1-399 (formerly TTP399)
- GK1-399, high dose, once per day (Experimental)
  Interventions: Drug: GK1-399 (formerly TTP399)
- GK1-399, high dose, twice per day (Experimental)
  Interventions: Drug: GK1-399 (formerly TTP399)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GK1-399 (formerly TTP399) — Treatment A: GK1-399 200 mg. Oral administration, twice per day.
  Arms: GK1-399, low dose
Drug: GK1-399 (formerly TTP399) — Treatment B: GK1-399 800 mg. Oral administration, once per day.
  Arms: GK1-399, high dose, once per day
Drug: GK1-399 (formerly TTP399) — Treatment C: GK1-399 800 mg. Oral administration, twice per day.
  Arms: GK1-399, high dose, twice per day
Drug: Placebo — Dose-matched placebo. Oral administration.
  Arms: Placebo

SUMMARY:
The purpose of this trial is to study the drug levels and biomarkers in the body and the safety of an investigational drug (GK1-399) in patients with Type 2 diabetes. Patients in the study will receive placebo for 1 week followed by 1 of 4 treatments for 6 weeks. One of the 4 treatments will be placebo, which does not contain an active ingredient. The study participation includes in-patient and out-patient days.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, aged 18 through 75 years at screening.
* Have a diagnosis of Type 2 Diabetes Mellitus (T2DM)
* On a stable dose of background medication for the treatment of diabetes
* Body Mass Index (BMI) between 20-40 kg/m2 (inclusive)

Exclusion Criteria:

* Subjects with type 1 diabetes, heart attack or stroke in the past 6 months, uncontrolled blood pressure, significant kidney disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of GK1-399 from plasma concentrations | 52 time points over a 6 week period
  Area under the plasma concentration verses time curve from time 0 to the end of the dosing interval, maximum plasma concentration

SECONDARY OUTCOMES:
Pharmacodynamic parameters of plasma glucose | 52 time points over a 6 week period
  Fasting plasma glucose and postprandial plasma glucose

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Burstein, Pharm.D., Study Director — TransTech Pharma, Inc.
Locations (11):
- United States (11):
  - Forest Investigative Site 009, Little Rock, Arkansas
  - Forest Investigative Site 006, Chula Vista, California
  - Forest Investigative Site 002, DeLand, Florida
  - Forest Investigative Site 001, Miami, Florida
  - Forest Investigative Site 010, Overland Park, Kansas
  - Forest Investigative site 011, Saint Paul, Minnesota
  - Forest Investigative Site 005, Springfield, Missouri
  - Forest Investigative Site 003, Neptune City, New Jersey
  - Forest Investigative Site 008, Willingboro, New Jersey
  - Forest Investigative Site 007, New York, New York
  - Forest Investigative Site 004, San Antonio, Texas